CLINICAL TRIAL: NCT02851407
Title: A Phase 3, Randomized, Adaptive Study Comparing the Efficacy and Safety of Defibrotide vs Best Supportive Care in the Prevention of Hepatic Veno-Occlusive Disease in Adult and Pediatric Patients Undergoing Hematopoietic Stem Cell Transplant
Brief Title: Study Comparing Efficacy and Safety of Defibrotide vs Best Supportive Care in the Prevention of Hepatic Veno-Occlusive Disease in Adult and Pediatric Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Jazz Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 15-007
Record Dates: First submitted 2016-07-27; First posted 2016-08-01 (Estimated); Results first posted 2022-03-02 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-02

CONDITIONS: Veno-occlusive Disease
Keywords: stem cell transplant; hematopoietic stem cell transplant (HSCT); veno-occlusive disease (VOD); sinusoidal obstruction syndrome (SOS)
MeSH Terms: conditions — Hepatic Veno-Occlusive Disease | interventions — defibrotide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Defibrotide (Experimental): Defibrotide is administered intravenously at a dose of 25 mg/kg/day in addition to best supportive care on the day before the first day of the conditioning regimen and will continue (for those patients without a VOD diagnosis) for a recommended minimum of 21 days and end no later than Day +30 post HSCT
  Interventions: Drug: Defibrotide
- Best Supportive Care (Other): Best supportive care alone (without the addition of defibrotide) according to institutional guidelines and patient need, is administered on the first day of conditioning and will continue until Day +30 post HSCT or hospital discharge, whichever is sooner, or diagnosis of VOD, if applicable
  Interventions: Other: Best Supportive Care

INTERVENTIONS:
Drug: Defibrotide
  Arms: Defibrotide
Other: Best Supportive Care
  Arms: Best Supportive Care

SUMMARY:
This study is to compare the efficacy and safety of defibrotide prophylaxis in addition to best supportive care versus best supportive care alone in the prevention of hepatic veno- occlusive disease (VOD) in adult and pediatric patients undergoing hematopoietic stem cell transplant who are at high risk or very high risk of developing VOD.

ELIGIBILITY:
Inclusion Criteria:

1. Patient must be above the age of 1 month as of the start date of study treatment.
2. Patient must be scheduled to undergo allogeneic hematopoietic stem cell transplant (HSCT) (adults or pediatric patients) or autologous HSCT (pediatric patients only) and be at high risk or very high risk of developing veno-occlusive disease (VOD).
3. Female patients (and female partners of male patients) of childbearing potential who are sexually active must agree to use a highly effective method of contraception with their partners during exposure to defibrotide and for 1 week after the last dose of defibrotide.
4. Adult patients must be able to understand and sign a written informed consent. For minor patients, the parent/legal guardian or representative must be able to understand and sign a written informed consent. Assent, when appropriate, will be obtained according to institutional guidelines.

Exclusion Criteria:

1. Patient has hemodynamic instability within 24 hours before the start of study treatment.
2. Patient has acute bleeding that is clinically significant within 24 hours before the start of study treatment.
3. Patient used any medication that increases the risk of bleeding within 24 hours before the start of study treatment.
4. Patient is using or plans to use an investigational agent for the prevention or treatment of VOD.
5. Patient, in the opinion of the investigator, may not be able to comply with the safety monitoring requirements of the study.
6. Patient or parent/legal guardian or representative has a psychiatric illness that would prevent the patient or parent/legal guardian or representative from giving informed consent and/or assent.
7. Patient has a serious active disease or co-morbid medical condition, as judged by the investigator, which would interfere with the conduct of this study.
8. Patient is pregnant or lactating and does not agree to stop breastfeeding.
9. Patient has a known history of hypersensitivity to defibrotide or any of the excipients.
10. Patient or parent/legal guardian or representative lacks the full mental capacity to understand and sign a written informed consent.
11. Patient is receiving or plans to receive other investigational therapy during study.

Min Age: 1 Month | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 372 (Actual)
Dates: Start 2016-09-01 (Actual); Primary Completion 2020-10-20 (Actual); Study Completion 2020-10-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jazz Pharmaceuticals, Study Director — Jazz Pharmaceuticals
Locations (114):
- United States (37):
  - Children's Hospital of Alabama, Birmingham, Alabama
  - Phoenix Children's Hospital, Phoenix, Arizona
  - University of Arizona Cancer Center, Tucson, Arizona
  - Children's Hospital Los Angeles, Los Angeles, California
  - Stanford University, Palo Alto, California
  - Rady Childrens Hospital San Diego, San Diego, California
  - University of California San Francisco, San Francisco, California
  - Colorado Children's Hospital, Aurora, Colorado
  - Alfred I Dupont Hospital For Children, Wilmington, Delaware
  - Nicklaus Childrens Hospital, Miami, Florida
  - Johns Hopkins All Children's Hospital, St. Petersburg, Florida
  - Children's Healthcare of Atlanta, Atlanta, Georgia
  - Ann and Robert H Lurie Childrens Hospital of Chicago, Chicago, Illinois
  - Tufts Floating Hospital for Children, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Children's Hospital of Michigan, Detroit, Michigan
  - Children's Mercy Hospital, Kansas City, Missouri
  - Columbia University Medical Center, New York, New York
  - Weill Cornell Medical College, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Children's Hospital at Montefiore, The Bronx, New York
  - Duke University Medical Center, Durham, North Carolina
  - University Hospital Case Medical Center, Cleveland, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Doernbecher Children's Hospital, Portland, Oregon
  - Penn State Milton S Hershey Medical Center, Hershey, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Medical University of South Carolina - PPDS, Charleston, South Carolina
  - Vanderbilt Ingram Cancer Center, Nashville, Tennessee
  - Children's Medical Center Dallas, Dallas, Texas
  - Cook Childrens Hospital, Fort Worth, Texas
  - MD Anderson Cancer Center, Houston, Texas
  - Texas Childrens Hospital, Houston, Texas
  - Primary Children's Hospital, Salt Lake City, Utah
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin
- Australia (2):
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Royal Children's Hospital Melbourne, Melbourne, Victoria
- Belgium (5):
  - Cliniques Universitaires Saint-Luc, Brussels
  - UZ Gent, Ghent
  - UZ Leuven Gasthuisberg, Leuven
  - UZ Leuven, Leuven
  - Centre Hospitalier Universitaire du Sart Tilman, Liège
- Canada (2):
  - Alberta Children's Hospital, Calgary, Alberta
  - Sainte Justine Hospital, Montreal, Quebec
- France (5):
  - Hopital Jean Minjoz, Besançon
  - Institut Paoli Calmettes, Marseille
  - Hôpital Saint Antoine, Paris
  - CHU de Poitiers, Poitiers
  - Institut Universitaire du Cancer de Toulouse - Oncopôle, Toulouse
- Germany (7):
  - Klinikum Frankfurt Oder GmbH, Frankfurt (Oder), Brandenburg
  - Universitätsklinikum der RWTH Aachen, Aachen, North Rhine-Westphalia
  - Universitätsklinikum Münster, Münster, North Rhine-Westphalia
  - Universitätsklinikum Carl Gustav Carus an der TU Dresden, Dresden, Saxony
  - Universitätsklinikum Leipzig, Leipzig, Saxony
  - Universitätsklinikum Hamburg Eppendorf, Hamburg
  - Klinikum der Universitat Regensburg, Regensburg
- Israel (6):
  - Rambam Health Care Campus, Haifa
  - Rambam Health Corporation, Haifa
  - Hadassah Ein Kerem Hospital, Jerusalem
  - Schneider Children Medical Center of Israel, Petah Tikva
  - Chaim Sheba Medical Center, Ramat Gan
  - Tel Aviv Sourasky Medical Center, Tel Aviv
- Italy (6):
  - 11. Azienda Ospedaliero Universitaria Ospedali Riuniti di Ancona-Umberto I G M Lancisi G Salesi, Ancona
  - Azienda Ospedaliero - Universitaria, Catania
  - Azienda Ospedaliera Universitaria Careggi, Florence
  - AORMN Marche Nord, Pesaro
  - Ospedale Pediatrico Bambino Gesù, Roma
  - Fondazione Policlinico Universitario A Gemelli, Roma
- Japan (14):
  - Anjo Kosei Hospital, Anjo
  - Hamanomachi Hospital, Fukuoka
  - Fukushima Medical University Hospital, Fukushima
  - Kobe University Hospital, Hyōgo
  - Kanagawa Children's Medical Center, Kanagawa
  - National Hospital Organization Kumamoto Medical Center, Kumamoto
  - Japanese Red Cross Nagoya Daiichi Hospital, Nagoya
  - Hyogo College of Medicine, Nishinomiya
  - Osaka International Cancer Institute, Osaka
  - Osaka City University Hospital, Osaka
  - Hokkaido University Hospital, Sapporo
  - Toranomon Hospital, Tokyo
  - Tokyo Metropolitan Cancer and Infectious Diseases Center Komagome Hospital, Tokyo
  - Medical Hospital Tokyo Medical and Dental University, Tokyo
- Auckland City Hospital, Auckland, New Zealand
- South Korea (5):
  - Seoul National University Hospital, Seoul
  - Severance Hospital at Yonsei University Health System, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - The Catholic University of Korea Seoul St. Mary's Hospital, Seoul
- Spain (11):
  - Hospital Universitario Germans Trias i Pujol, Badalona, Barcelona
  - Hospital Universitario Vall d Hebron, Barcelona
  - Hospital Universitario Reina Sofia, Córdoba
  - Hospital Sant Joan de Deu - PIN, Esplugues de Llobregat
  - Hospital Infantil Universitario Niño Jesus, Madrid
  - Hospital Universitario Ramon y Cajal, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Regional Universitario de Malaga Hospital General, Málaga
  - Hospital General Universitario Morales Meseguer, Murcia
  - Hospital Universitario de Salamanca, Salamanca
  - Hospital Universitario Virgen del Rocio, Seville
- Turkey (Türkiye) (7):
  - Akdeniz University Medical Faculty Department of Pediatrics, Antalya, Konyaalti
  - Erciyes University Medical Faculty, Kayseri, Talas
  - Medicana International Ankara Hospital, Ankara
  - Medical Park Antalya Hospital, Antalya
  - Ege Universitesi Tip Fakultesi, Bornova
  - Acibadem Universitesi Tip Fakultesi Atakent Hastanesi, Istanbul
  - Acibadem Adana Hospital, Seyhan
- United Kingdom (6):
  - Birmingham Children's Hospital, Birmingham
  - Beatson West of Scotland Cancer Centre, Glasgow
  - Royal Hospital for Children, Glasgow
  - St. James University Hospital, Leeds
  - Kings College Hospital, London
  - Great Ormond Street Hospital, London

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Corbacioglu S, Grupp SA, Richardson PG, Duarte R, Pagliuca A, Ruutu T, Mahadeo K, Carreras E. Prevention of veno-occlusive disease/sinusoidal obstruction syndrome: a never-ending story and no easy answer. Bone Marrow Transplant. 2023 Aug;58(8):839-841. doi: 10.1038/s41409-023-02007-2. Epub 2023 May 25. No abstract available. PMID 37231094
- [Derived] Grupp SA, Corbacioglu S, Kang HJ, Teshima T, Khaw SL, Locatelli F, Maertens J, Stelljes M, Stepensky P, Lopez P, Amber V, Pagliuca A, Richardson PG, Mohty M. Defibrotide plus best standard of care compared with best standard of care alone for the prevention of sinusoidal obstruction syndrome (HARMONY): a randomised, multicentre, phase 3 trial. Lancet Haematol. 2023 May;10(5):e333-e345. doi: 10.1016/S2352-3026(23)00011-X. Epub 2023 Mar 28. PMID 37001534

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants, their parents/legal guardians, or representatives were required to sign a statement of informed consent.
Groups:
- Defibrotide Prophylaxis: Defibrotide was administered intravenously at a dose of 6.25mg/kg/day in 4 divided doses by IV infusion over 2 hours in addition to best supportive care within 24 hours before the first dose of the conditioning regimen and continued (for those participants without a VOD diagnosis) for a recommended minimum of 21 days and end no later than Day +30 post-HSCT.
- Best Supportive Care: Best supportive care alone (without the addition of defibrotide) according to institutional guidelines and participant need, was administered on the first day of conditioning and continued until Day +30 post HSCT or hospital discharge, whichever was sooner, or diagnosis of VOD, if applicable.
Period: Overall Study
Arm/Group | Defibrotide Prophylaxis | Best Supportive Care
Started | 190 | 182
Completed | 120 | 121
Not Completed | 70 | 61
Not completed — Withdrawal by parent/guardian | 2 | 7
Not completed — Protocol deviation | 0 | 1
Not completed — Transferred to another hospital to continue | 1 | 0
Not completed — Other Death | 30 | 20
Not completed — Adverse event, serious fatal | 6 | 8
Not completed — Consent withdrawn by participant | 5 | 3
Not completed — Screen failure | 2 | 1
Not completed — Disease relapse | 9 | 6
Not completed — Physician Decision | 7 | 6
Not completed — Transferred to hospital closer to home | 0 | 1
Not completed — Enrolled in an investigational study | 0 | 1
Not completed — Early recovery | 1 | 0
Not completed — Adverse event, non-fatal | 7 | 5
Not completed — Lost to Follow-up | 0 | 2

BASELINE CHARACTERISTICS:
Population: Baseline characteristics were assessed using the Intent-to-Treat Analysis Set.
Groups:
- Best Supportive Care: Best supportive care alone (without the addition of defibrotide) according to institutional guidelines and participant need, was administered on the first day of conditioning and continued until Day +30 post HSCT or hospital discharge, whichever was sooner, or diagnosis of VOD, if applicable.
  Best Supportive Care
- Total: Total of all reporting groups
Arm/Group | Defibrotide Prophylaxis | Best Supportive Care | Total
Number analyzed (Participants) | 190 | 182 | 372
Age, Continuous [Mean (Standard Deviation); unit: years] | 22.7 (21.87) | 23.2 (21.73) | 23.0 (21.77)
Age, Customized [Count of Participants; unit: Participants]
  Participants ≤16 Years | 104 | 94 | 198
  Participants >16 Years | 86 | 88 | 174
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 90 | 82 | 172
  Male | 100 | 100 | 200
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 22 | 21 | 43
  Not Hispanic or Latino | 150 | 143 | 293
  Unknown or Not Reported | 18 | 18 | 36
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 39 | 46 | 85
  Native Hawaiian or Other Pacific Islander | 0 | 2 | 2
  Black or African American | 5 | 8 | 13
  White | 125 | 109 | 234
  More than one race | 2 | 0 | 2
  Unknown or Not Reported | 19 | 17 | 36

OUTCOME MEASURES:

1. Primary Outcome: Veno-occlusive Disease (VOD)-Free Survival by Day +30 Post-Hematopoietic Stem Cell Transplant (HSCT) Per the Independent Endpoint Adjudication Committee (EPAC)
Description: VOD-free survival is a composite of survival status and VOD occurrence as determined by modified Seattle criteria adjudicated by a blinded independent EPAC. An event is defined as a VOD diagnosis (as assessed by the EPAC) or death, whichever, is earlier, up to and including Day +30 post-HSCT. The values reported below are participants who did not experience VOD or death by Day +30 post-HSCT.
Time Frame: Day +30 Post-HSCT
Population: VOD-free survival was assessed using the Intent-to-Treat Analysis Set.
Measure: Number (95% Confidence Interval); unit: KM Estimate % of participants
Arm/Group | Defibrotide Prophylaxis | Best Supportive Care
Number analyzed (Participants) | 190 | 182
KM Estimate % of participants | 66.8 [57.8 to 74.4] | 72.5 [62.3 to 80.4]

2. Secondary Outcome: Veno-Occlusive Disease (VOD)-Free Survival by Day +100 Post-Hematopoietic Stem Cell Transplant (HSCT) Per the Independent Endpoint Adjudication Committee (EPAC)
Description: VOD-free survival is a composite of survival status and VOD occurrence as determined by modified Seattle criteria adjudicated by a blinded independent EPAC. An event is defined as a VOD diagnosis (as assessed by the EPAC) or death, whichever, is earlier, up to and including Day +100 post-HSCT. The values reported below are participants who did not experience VOD or death by Day +100 post-HSCT.
Time Frame: Day +100 Post-HSCT
Population: VOD-free survival was assessed using the Intent-to-Treat Analysis Set.
Measure: Number (95% Confidence Interval); unit: KM Estimate % of participants
Arm/Group | Defibrotide Prophylaxis | Best Supportive Care
Number analyzed (Participants) | 190 | 182
KM Estimate % of participants | 49.8 [26.1 to 69.5] | 57.1 [36.6 to 73.1]

3. Secondary Outcome: Percentage of Participants With Veno-Occlusive Disease (VOD) by Day +30 Post-Hematopoietic Stem Cell Transplant (HSCT)
Description: The number of participants who were diagnosed with VOD based on the Modified Seattle Criteria as per blinded EPAC assessment. The percentage was calculated out of the total number of participants in each arm of the study. The values reported below are the numbers and percentages of participants who experienced VOD by Day +30 post-HSCT.
Time Frame: Day +30 Post-HSCT
Population: Percentage of Participants with VOD by Day +30 post-HSCT was assessed using the Intent-to-Treat Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | Defibrotide Prophylaxis | Best Supportive Care
Number analyzed (Participants) | 190 | 182
Participants | 47 | 38

4. Secondary Outcome: Veno-Occlusive Disease (VOD)-Free Survival Rate by Day +180 Post-Hematopoietic Stem Cell Transplant (HSCT)
Description: VOD-free survival is a composite of survival status and VOD occurrence as determined by modified Seattle criteria. An event is defined as a VOD diagnosis or death, whichever, is earlier, up to and including Day +180 post-HSCT. The diagnosis of VOD through Day +100 post-HSCT was based on Endpoint Adjudication Committee (EPAC), and the diagnosis of VOD after Day +100 post-HSCT was based on investigator assessments. The values reported below are participants who did not experience VOD or death by Day +180 post-HSCT.
Time Frame: Day +180 Post-HSCT
Population: VOD-free Survival by Day +180 post-HSCT was assessed using the Intent-to-Treat Analysis Set.
Measure: Number (95% Confidence Interval); unit: KM Estimate % of participants
Arm/Group | Defibrotide Prophylaxis | Best Supportive Care
Number analyzed (Participants) | 190 | 182
KM Estimate % of participants | 34.6 [18.2 to 51.8] | 42.8 [26.7 to 58.0]

5. Secondary Outcome: Non-Relapse Mortality (NRM) for Defibrotide (DP) and Best Supportive Care (BSC) by Days +100 and +180 Post-Hematopoietic Stem Cell Transplant (HSCT)
Description: NRM is defined as death that occurs after HSCT in participants who were noted as having malignant primary disease on the disease history electronic case report form (eCRF) and do not have primary disease relapse post-HSCT.
Time Frame: Days +100 and +180 Post-HSCT
Population: Non-relapse mortality was assessed using the number of participants with malignant primary disease within treatment arm from the Intent-to-Treat Analysis Set.
Measure: Number (95% Confidence Interval); unit: KM Estimate % of non-relapse survival
Arm/Group | Defibrotide Prophylaxis | Best Supportive Care
Number analyzed (Participants) | 147 | 139
KM Estimate % of non-relapse survival
  Day +100 Post-HSCT | 80.4 [71.6 to 86.8] | 89.7 [82.1 to 94.2]
  Day +180 Post-HSCT | 77.9 [68.4 to 84.9] | 81.9 [70.8 to 89.1]

6. Secondary Outcome: Percentage of Participants With Veno-Occlusive Disease (VOD)-Associated Multi-Organ Dysfunction (MOD) by Days +30 and Days +100 Post-Hematopoietic Stem Cell Transplant (HSCT) in Patients Who Developed VOD
Description: VOD-associated MOD is defined for participants as occurring if the investigator answers "Yes" to the question "Has the participant been diagnosed with VOD associated MOD?" in the electronic case report form (eCRF). The values below are the number of participants who received the answer, "Yes."
Time Frame: Days +30 and +100 Post-HSCT
Population: Percentage of Participants with VOD-associated MOD was assessed using the Intent-to-Treat Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | Defibrotide Prophylaxis | Best Supportive Care
Number analyzed (Participants) | 190 | 182
Participants
  Day +30 Post-HSCT | 8 | 8
  Day +100 Post-HSCT | 9 | 10

7. Secondary Outcome: Percentage of Participants Who Had Resolution of Veno-Occlusive Disease (VOD) by Day +180 Post-Hematopoietic Stem Cell Transplant (HSCT)
Description: The proportion of participants who had resolution of VOD by Day +180 post-HSCT is reported as a percentage.
Time Frame: Day +180 Post-HSCT
Population: Resolution of VOD was assessed using the Intent-To-Treat Analysis Set. The overall number analyzed is the number of participants diagnosed with VOD by Day +30 post-HSCT by the investigator.
Measure: Count of Participants; unit: Participants
Arm/Group | Defibrotide Prophylaxis | Best Supportive Care
Number analyzed (Participants) | 23 | 29
Participants | 6 | 15

8. Secondary Outcome: Time to Resolution of Veno-Occlusive Disease (VOD) by Day +180 Post-Hematopoietic Stem Cell Transplant (HSCT)
Description: Time to Resolution of VOD is calculated as follows: Time to Resolution of VOD= [Date of VOD resolution] - [Date of VOD diagnosis by investigator].
Time Frame: Day +180 Post-HSCT
Population: Resolution of VOD was assessed using the Intent-To-Treat Analysis.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Defibrotide Prophylaxis | Best Supportive Care
Number analyzed (Participants) | 190 | 182
Days | NA [NA to NA] — Not assessable. There were not enough participants who had VOD resolution for this to be estimated. The value is not estimable because the number of VOD resolution, i.e 6, is less than half of the number of diagnosed VOD in the DP arm, so the KM estimate of median time cannot be evaluated. | 30.0 [21.0 to 48.0]

9. Secondary Outcome: Percentage of Participants With Veno-Occlusive Disease (VOD) After Day +30 Post-Hematopoietic Stem Cell Transplant (HSCT) up to Days +100 and +180 Post-HSCT
Description: The values shown are the number and percentage of participants with VOD after day +30 post-HSCT and on or before Days +100 and +180 post-HSCT. The diagnosis of VOD through Day +100 post-HSCT was made by Endpoint Adjudication Committee (EPAC), and the diagnosis of VOD after Day +100 post-HSCT was based on investigator assessments.
Time Frame: Days +100 and +180 Post-HSCT
Population: Percentage of VOD was assessed using the Intent-to-Treat Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | Defibrotide Prophylaxis | Best Supportive Care
Number analyzed (Participants) | 190 | 182
Participants
  Day +100 Post-HSCT | 6 | 5
  Day +180 Post-HSCT | 6 | 5

10. Secondary Outcome: Change in 5-Level EuroQol-5D (EQ-5D-5L) Dimensions From Baseline to Day +180 Post-Hematopoietic Stem Cell Transplant (HSCT) for Adult Participants Age ≥ 16 Years: Mobility
Description: For each of the five dimensions of mobility, self-care, activity, pain, and anxiety based on the descriptive system of the EQ-5D-5L, the numbers and percentages of participants for all categories (the three levels of reported problems and question not completed) at Day +180 Post-HSCT was assessed. Each dimension was categorized as follows: Condition improved, if the reported level of problem is lower at the assessment than baseline; condition unchanged, if the reported level of problem remains the same; condition deteriorated, if the reported level of problem is higher at that assessment than at baseline; and unknown, if the reported level of problem is missing either at baseline or at that assessment.
Time Frame: Day +180 Post-HSCT
Population: EQ-5D-5L Mobility was assessed using the Age ≥ 16 Years Safety Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | Defibrotide Prophylaxis | Best Supportive Care
Number analyzed (Participants) | 45 | 46
Participants
  Condition improved | 4 | 7
  Condition unchaged | 28 | 28
  Condition deteriorated | 9 | 6
  Unknown | 4 | 5

11. Secondary Outcome: Change in 5-Level EuroQol-5D (EQ-5D-5L) Dimensions From Baseline to Day +180 Post-Hematopoietic Stem Cell Transplant (HSCT) for Adult Participants Age ≥ 16 Years: Self-Care
Description: as for outcome 10
Time Frame: Day +180 Post-HSCT
Population: EQ-5D-5L Self-Care was assessed using the Age ≥ 16 Years Safety Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | Defibrotide Prophylaxis | Best Supportive Care
Number analyzed (Participants) | 45 | 46
Participants
  Condition improved | 3 | 6
  Condition unchaged | 35 | 32
  Condition deteriorated | 3 | 4
  Unknown | 4 | 4

12. Secondary Outcome: Change in 5-Level EuroQol-5D (EQ-5D-5L) Dimensions From Baseline to Day +180 Post-Hematopoietic Stem Cell Transplant (HSCT) for Adult Participants Age ≥ 16 Years: Activity
Description: as for outcome 10
Time Frame: Day +180 Post-HSCT
Population: EQ-5D-5L Activity was assessed using the Age ≥ 16 Years Safety Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | Defibrotide Prophylaxis | Best Supportive Care
Number analyzed (Participants) | 45 | 46
Participants
  Condition improved | 7 | 10
  Condition unchaged | 24 | 22
  Condition deteriorated | 9 | 10
  Unknown | 5 | 4

13. Secondary Outcome: Change in 5-Level EuroQol-5D (EQ-5D-5L) Dimensions From Baseline to Day +180 Post-Hematopoietic Stem Cell Transplant (HSCT) for Adult Participants Age ≥ 16 Years: Pain
Description: as for outcome 10
Time Frame: Day +180 Post-HSCT
Population: EQ-5D-5L Pain was assessed using the Age ≥ 16 Years Safety Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | Defibrotide Prophylaxis | Best Supportive Care
Number analyzed (Participants) | 45 | 46
Participants
  Condition improved | 10 | 11
  Condition unchaged | 25 | 19
  Condition deteriorated | 6 | 12
  Unknown | 4 | 4

14. Secondary Outcome: Change in 5-Level EuroQol-5D (EQ-5D-5L) Dimensions From Baseline to Day +180 Post-Hematopoietic Stem Cell Transplant (HSCT) for Adult Participants Age ≥ 16 Years: Anxiety
Description: as for outcome 10
Time Frame: Day +180 Post-HSCT
Population: EQ-5D-5L Anxiety was assessed using the Age ≥ 16 Years Safety Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | Defibrotide Prophylaxis | Best Supportive Care
Number analyzed (Participants) | 45 | 46
Participants
  Condition improved | 11 | 11
  Condition unchaged | 22 | 27
  Condition deteriorated | 7 | 4
  Unknown | 5 | 4

15. Secondary Outcome: Change in EuroQol-5D for Youth (EQ-5D-Y) Dimensions From Baseline to Day +180 Post-Hematopoietic Stem Cell Transplant (HSCT) for Pediatric Participants Age ≥ 4 and ≤ 7 Years: Mobility
Description: For each of the five dimensions of mobility, self-care, activity, pain, and anxiety based on the descriptive system of the EQ-5D-Y, self-report version, the numbers and percentages of participants for all categories (the three levels of reported problems and question not completed) at Day +180 post-HSCT was assessed. Each dimension was categorized as follows: Condition improved, if the reported level of problem is lower at the assessment than baseline; condition unchanged, if the reported level of problem remains the same; condition deteriorated, if the reported level of problem is higher at that assessment than at baseline; and unknown, if the reported level of problem is missing either at baseline or at that assessment.
Time Frame: Day +180 Post-HSCT
Population: EQ-5D-Y Mobility was assessed using the Age ≥ 4 and ≤ 7 Years Safety Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | Defibrotide Prophylaxis | Best Supportive Care
Number analyzed (Participants) | 15 | 15
Participants
  Condition improved | 2 | 1
  Condition unchanged | 8 | 8
  Condition deteriorated | 3 | 4
  Unknown | 2 | 2

16. Secondary Outcome: Change in EuroQol-5D for Youth (EQ-5D-Y) Dimensions From Baseline to Day +180 Post-Hematopoietic Stem Cell Transplant (HSCT) for Pediatric Participants Age ≥ 4 and ≤ 7 Years: Self-Care
Description: as for outcome 15
Time Frame: Day +180 Post-HSCT
Population: EQ-5D-Y Self-Care was assessed using the Age ≥ 4 and ≤ 7 Years Safety Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | Defibrotide Prophylaxis | Best Supportive Care
Number analyzed (Participants) | 15 | 15
Participants
  Condition improved | 3 | 2
  Condition unchanged | 7 | 10
  Condition deteriorated | 3 | 1
  Unknown | 2 | 2

17. Secondary Outcome: Change in EuroQol-5D for Youth (EQ-5D-Y) Dimensions From Baseline to Day +180 Post-Hematopoietic Stem Cell Transplant (HSCT) for Pediatric Participants Age ≥ 4 and ≤ 7 Years: Activity
Description: as for outcome 15
Time Frame: Day +180 Post-HSCT
Population: EQ-5D-Y Activity was assessed using the Age ≥ 4 and ≤ 7 Years Safety Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | Defibrotide Prophylaxis | Best Supportive Care
Number analyzed (Participants) | 15 | 15
Participants
  Condition improved | 2 | 1
  Condition unchanged | 7 | 11
  Condition deteriorated | 4 | 1
  Unknown | 2 | 2

18. Secondary Outcome: Change in EuroQol-5D for Youth (EQ-5D-Y) Dimensions From Baseline to Day +180 Post-Hematopoietic Stem Cell Transplant (HSCT) for Pediatric Participants Age ≥ 4 and ≤ 7 Years: Pain
Description: as for outcome 15
Time Frame: Day +180 Post-HSCT
Population: EQ-5D-Y Pain was assessed using the Age ≥ 4 and ≤ 7 Years Safety Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | Defibrotide Prophylaxis | Best Supportive Care
Number analyzed (Participants) | 15 | 15
Participants
  Condition improved | 4 | 3
  Condition unchanged | 7 | 9
  Condition deteriorated | 2 | 1
  Unknown | 2 | 2

19. Secondary Outcome: Change in EuroQol-5D for Youth (EQ-5D-Y) Dimensions From Baseline to Day +180 Post-Hematopoietic Stem Cell Transplant (HSCT) for Pediatric Participants Age ≥ 4 and ≤ 7 Years: Anxiety
Description: as for outcome 15
Time Frame: Day +180 Post-HSCT
Population: EQ-5D-Y Anxiety was assessed using the Age ≥ 4 and ≤ 7 Years Safety Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | Defibrotide Prophylaxis | Best Supportive Care
Number analyzed (Participants) | 15 | 15
Participants
  Condition improved | 3 | 2
  Condition unchanged | 8 | 10
  Condition deteriorated | 2 | 1
  Unknown | 2 | 2

20. Secondary Outcome: Change in EuroQol-5D for Youth (EQ-5D-Y) Dimensions From Baseline to Day +180 Post-Hematopoietic Stem Cell Transplant (HSCT) for Pediatric Participants Age ≥ 8 and ≤ 15 Years: Mobility
Description: as for outcome 15
Time Frame: Day +180 Post-HSCT
Population: EQ-5D-Y Mobility at Day +180 post-HSCT was assessed using participants Age ≥ 8 and ≤ 15 Years Safety Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | Defibrotide Prophylaxis | Best Supportive Care
Number analyzed (Participants) | 14 | 17
Participants
  Condition improved | 1 | 2
  Condition unchanged | 9 | 10
  Condition deteriorated | 3 | 4
  unknown | 1 | 1

21. Secondary Outcome: Change in EuroQol-5D for Youth (EQ-5D-Y) Dimensions From Baseline to Day +180 Post-Hematopoietic Stem Cell Transplant (HSCT) for Pediatric Participants Age ≥ 8 and ≤ 15 Years: Self-Care
Description: as for outcome 15
Time Frame: Day +180 Post-HSCT
Population: EQ-5D-Y Self-Care at Day +180 post-HSCT was assessed using participants Age ≥ 8 and ≤ 15 Years Safety Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | Defibrotide Prophylaxis | Best Supportive Care
Number analyzed (Participants) | 14 | 17
Participants
  Condition improved | 3 | 4
  Condition unchanged | 8 | 10
  Condition deteriorated | 2 | 2
  Unknown | 1 | 1

22. Secondary Outcome: Change in EuroQol-5D for Youth (EQ-5D-Y) Dimensions From Baseline to Day +180 Post-Hematopoietic Stem Cell Transplant (HSCT) for Pediatric Participants Age ≥ 8 and ≤ 15 Years: Activity
Description: as for outcome 15
Time Frame: Day +180 Post-HSCT
Population: EQ-5D-Y Activity at Day +180 post-HSCT was assessed using participants Age ≥ 8 and ≤ 15 Years Safety Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | Defibrotide Prophylaxis | Best Supportive Care
Number analyzed (Participants) | 14 | 17
Participants
  Condition improved | 1 | 3
  Condition unchanged | 7 | 10
  Condition deteriorated | 5 | 3
  Unknown | 1 | 1

23. Secondary Outcome: Change in EuroQol-5D for Youth (EQ-5D-Y) Dimensions From Baseline to Day +180 Post-Hematopoietic Stem Cell Transplant (HSCT) for Pediatric Participants Age ≥ 8 and ≤ 15 Years: Pain
Description: as for outcome 15
Time Frame: Day +180 Post-HSCT
Population: EQ-5D-Y Pain at Day +180 post-HSCT was assessed using participants Age ≥ 8 and ≤ 15 Years Safety Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | Defibrotide Prophylaxis | Best Supportive Care
Number analyzed (Participants) | 14 | 17
Participants
  Condition improved | 0 | 5
  Condition unchanged | 12 | 8
  Condition deteriorated | 1 | 3
  Unknown | 1 | 1

24. Secondary Outcome: Change in EuroQol-5D for Youth (EQ-5D-Y) Dimensions From Baseline to Day +180 Post-Hematopoietic Stem Cell Transplant (HSCT) for Pediatric Participants Age ≥ 8 and ≤ 15 Years: Anxiety
Description: as for outcome 15
Time Frame: Day +180 Post-HSCT
Population: EQ-5D-Y Pain at Day +180 post-HSCT was assessed using participants Age ≥ 8 and ≤ 15 Years Safety Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | Defibrotide Prophylaxis | Best Supportive Care
Number analyzed (Participants) | 14 | 17
Participants
  Condition improved | 6 | 6
  Condition unchanged | 5 | 8
  Condition deteriorated | 2 | 2
  Unknown | 1 | 1

25. Secondary Outcome: Maximum Plasma Concentration (Cmax) of Defibrotide Prophylaxis During the Prophylaxis Phase
Description: Cmax is the maximum defibrotide plasma concentration, obtained directly from the observed data. Cmax is a summary statistic and it is not reported on an hourly basis. If veno-occlusive disease (VOD) occurs, the prophylaxis phase starts on the baseline date and ends on the day before the start date of rescue defibrotide. If VOD does not occur, the prophylaxis phase starts on the baseline date and ends on the date of study completion/early termination.
Time Frame: Day +1 and +7 Post-HSCT
Population: Cmax was assessed using the Pharmacokinetic (PK) Evaluable Analysis Set. Intensive PK samples were collected during the prophylaxis phase on Day +1 and Day +7 post-HSCT in a subgroup of participants in the DP arm who separately consented for this sampling. Sparse PK samples were collected from participants throughout the study according to the protocol.
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | Defibrotide Prophylaxis | Best Supportive Care
Number analyzed (Participants) | 2 | 0
μg/mL
  Day +1 Post-HSCT | 30.4 (10.600) |
  Day +7 Post-HSCT | 40 (3.168) |

26. Secondary Outcome: Area Under the Defibrotide Concentration-Time Curve (AUClast) of Defibrotide Prophylaxis During the Prophylaxis Phase
Description: AUClast is the area under the defibrotide concentration-time curve from 0 (pre-dose) to time of last quantifiable defibrotide concentration at time "t". AUClast is a summary statistic and it is not reported on an hourly basis. If veno-occlusive disease (VOD) occurs, the prophylaxis phase starts on the baseline date and ends on the day before the start date of rescue defibrotide. If VOD does not occur, the prophylaxis phase starts on the baseline date and ends on the date of study completion/early termination.
Time Frame: Day +1 and +7 Post-HSCT
Population: AUClast was assessed using the Pharmacokinetic (PK) Evaluable Analysis Set. Intensive PK samples were collected during the prophylaxis phase on Day +1 and Day +7 post-HSCT in a subgroup of participants in the DP arm who separately consented for this sampling. Sparse PK samples were collected from participants throughout the study according to the protocol.
Measure: Mean (Standard Deviation); unit: h*μg/mL
Arm/Group | Defibrotide Prophylaxis | Best Supportive Care
Number analyzed (Participants) | 2 | 0
h*μg/mL
  Day +1 Post-HSCT | 61.6 (28.488) |
  Day +7 Post-HSCT | 78.2 (10.781) |

27. Secondary Outcome: Mean Clearance of Defibrotide Prophylaxis During the Prophylaxis Phase
Description: Mean systemic clearance after intravenous dosing. Mean clearance is a summary statistic and it is not reported on an hourly basis. If veno-occlusive disease (VOD) occurs, the prophylaxis phase starts on the baseline date and ends on the day before the start date of rescue defibrotide. If VOD does not occur, the prophylaxis phase starts on the baseline date and ends on the date of study completion/early termination.
Time Frame: Day +1 and +7 Post-HSCT
Population: Mean clearance was assessed using the Pharmacokinetic (PK) Evaluable Analysis Set. Intensive PK samples were collected during the prophylaxis phase on Day +1 and Day +7 post-HSCT in a subgroup of participants in the DP arm who separately consented for this sampling. Sparse PK samples were collected from participants throughout the study according to the protocol.
Measure: Mean (Standard Deviation); unit: L/h
Arm/Group | Defibrotide Prophylaxis | Best Supportive Care
Number analyzed (Participants) | 2 | 0
L/h
  Day +1 Post-HSCT | 4.7 (0.304) |
  Day +7 Post-HSCT: number analyzed (Participants) | 0 | 0

28. Secondary Outcome: Volume of Distribution of Defibrotide Prophylaxis During the Prophylaxis Phase
Description: Mean volume of distribution following intravenous dosing. Mean volume of distribution is a summary statistic and it is not reported on an hourly basis.If veno-occlusive disease (VOD) occurs, the prophylaxis phase starts on the baseline date and ends on the day before the start date of rescue defibrotide. If VOD does not occur, the prophylaxis phase starts on the baseline date and ends on the date of study completion/early termination.
Time Frame: Day +1 and +7 Post-HSCT
Population: Volume of distribution was assessed using the Pharmacokinetic (PK) Evaluable Analysis Set. Intensive PK samples were collected during the prophylaxis phase on Day +1 and Day +7 post-HSCT in a subgroup of participants in the DP arm who separately consented for this sampling. Sparse PK samples were collected from participants throughout the study according to the protocol.
Measure: Mean (Standard Deviation); unit: L
Arm/Group | Defibrotide Prophylaxis | Best Supportive Care
Number analyzed (Participants) | 2 | 0
L
  Day +1 Post-HSCT | 7.9 (0.689) |
  Day +7 Post-HSCT | 5.9 (1.609) |

29. Secondary Outcome: Maximum Plasma Concentration (Cmax) of Defibrotide Prophylaxis During the Rescue Phase
Description: Cmax is the maximum defibrotide plasma concentration, obtained directly from the observed data. Cmax is a summary statistic and it is not reported on an hourly basis. For the subset of participants who developed veno-occlusive disease (VOD) and received rescue defibrotide, the rescue treatment phase begins on the start date of rescue defibrotide and ends on the date of study completion/early termination.
Time Frame: Day +14 Post-VOD Treatment
Population: Cmax was assessed using the Pharmacokinetic (PK) Evaluable Analysis Set. Frequent PK samples were collected from participants who developed VOD and received defibrotide rescue treatment (rescue phase) on VOD treatment Day 14. Sparse PK samples were collected from participants throughout the study according to the protocol.
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | Defibrotide Prophylaxis | Best Supportive Care
Number analyzed (Participants) | 4 | 14
μg/mL | 44.4 (18.550) | 39.7 (25.775)

30. Secondary Outcome: Area Under the Defibrotide Concentration-Time Curve (AUClast) of Defibrotide Prophylaxis During the Rescue Phase
Description: AUClast is the area under the defibrotide concentration-time curve from 0 (pre-dose) to time of last quantifiable defibrotide concentration at time "t". AUClast is a summary statistic and it is not reported on an hourly basis. For the subset of participants who developed veno-occlusive disease (VOD) and received rescue defibrotide, the rescue treatment phase begins on the start date of rescue defibrotide and ends on the date of study completion/early termination.
Time Frame: Day +14 Post-VOD Treatment
Population: AUClast was assessed using the Pharmacokinetic (PK) Evaluable Analysis Set. Frequent PK samples were collected from participants who developed VOD and received defibrotide rescue treatment (rescue phase) on VOD treatment Day 14. Sparse PK samples were collected from participants throughout the study according to the protocol.
Measure: Mean (Standard Deviation); unit: h*μg/mL
Arm/Group | Defibrotide Prophylaxis | Best Supportive Care
Number analyzed (Participants) | 4 | 14
h*μg/mL | 119.1 (68.875) | 90.7 (54.798)

31. Secondary Outcome: Volume of Distribution of Defibrotide Prophylaxis During the Rescue Phase
Description: Mean volume of distribution following intravenous dosing. Mean volume of distribution is a summary statistic and it is not reported on an hourly basis. For the subset of participants who developed veno-occlusive disease (VOD) and received rescue defibrotide, the rescue treatment phase begins on the start date of rescue defibrotide and ends on the date of study completion/early termination.
Time Frame: Day +14 Post-VOD Treatment
Population: Volume of distribution was assessed using the Pharmacokinetic (PK) Evaluable Analysis Set. Frequent PK samples were collected from participants who developed VOD and received defibrotide rescue treatment (rescue phase) on VOD treatment Day 14. Sparse PK samples were collected from participants throughout the study according to the protocol.
Measure: Mean (Standard Deviation); unit: L
Arm/Group | Defibrotide Prophylaxis | Best Supportive Care
Number analyzed (Participants) | 2 | 9
L | 6.3 (0.654) | 6.7 (5.895)

32. Secondary Outcome: Percentage of Participants With Grades 2, 3, and 4 Acute Graft-Versus-Host-Disease (GvHD) by Days +30, +100, and +180 Post-Hematopoietic Stem Cell Transplant (HSCT) in the Prophylaxis Phase
Description: The number and percentage of participants with Grade 2-4 acute GvHD in the prophylaxis phase. Grade 2 is defined as Skin stage = 3, or Liver stage = 1, or GI stage = 1. Grade 3 is defined as Skin stage = 3, or Liver stage = 2-3, or GI stage = 2-4. Grade 4 is defined as a Skin stage = 4, or Liver stage = 4, or GI stage = 2-4.
Time Frame: Days +30, +100, and +180 Post-HSCT
Population: Percentage of participants with acute GvHD was assessed using the Safety Analysis Set. Percentages were calculated with the number of participants in Safety Analysis Set who entered the study phase in each arm as a denominator during the prophylaxis phase.
Measure: Count of Participants; unit: Participants
Arm/Group | Defibrotide Prophylaxis | Best Supportive Care
Number analyzed (Participants) | 147 | 142
Participants
  Day +30 Post-HSCT | 13 | 13
  Day +100 Post-HSCT | 20 | 24
  Day +180 Post-HSCT | 22 | 26

33. Secondary Outcome: Percentage of Participants With Grades 2, 3, and 4 Acute Graft-Versus-Host-Disease (GvHD) by Days +30, +100, and +180 Post-Hematopoietic Stem Cell Transplant (HSCT) in the Rescue Phase
Description: The number and percentage of participants with Grade 2-4 acute GvHD in the rescue phase. Grade 2 is defined as Skin stage = 3, or Liver stage = 1, or GI stage = 1. Grade 3 is defined as Skin stage = 3, or Liver stage = 2-3, or GI stage = 2-4. Grade 4 is defined as a Skin stage = 4, or Liver stage = 4, or GI stage = 2-4.
Time Frame: Days +30, +100, and +180 Post-HSCT
Population: Percentage of participants with acute GvHD was assessed using the Safety Analysis Set. Percentages were calculated with the number of participants in Safety Analysis Set who entered the study phase in each arm as a denominator during the rescue phase.
Measure: Count of Participants; unit: Participants
Arm/Group | Defibrotide Prophylaxis | Best Supportive Care
Number analyzed (Participants) | 23 | 28
Participants
  Day +30 Post-HSCT | 5 | 1
  Day +100 Post-HSCT | 6 | 1
  Day +180 Post-HSCT | 6 | 1

34. Secondary Outcome: Percentage of Participants With Chronic Graft-Versus-Host-Disease (GvHD) by Day +180 Post-Hematopoietic Stem Cell Transplant (HSCT)
Description: The values shown are the number and percentages of participants who developed chronic GvHD by Day +180 post-HSCT in the prophylaxis phase and rescue phase.
Time Frame: Day +180 Post-HSCT
Population: Percentage of participants chronic GvHD was assessed using the Safety Analysis Set. Percentages were calculated with the number of participants in Safety Analysis Set who entered the study phase in each arm as a denominator. The number analyzed differs from the overall number of participants analyzed due to the count of participants included in the prophylaxis phase versus the rescue phase.
Measure: Count of Participants; unit: Participants
Arm/Group | Defibrotide Prophylaxis | Best Supportive Care
Number analyzed (Participants) | 181 | 174
Participants
  Prophylaxis Phase | 14 | 12
  Rescue Phase: number analyzed (Participants) | 23 | 28
  Rescue Phase | 2 | 1

35. Secondary Outcome: Number of Participants With Graft Failure During the Prophylaxis Phase and Rescue Phase
Description: Graft failure is defined as participants that after hematopoietic stem cell transplant (HSCT) never reached an absolute neutrophil count >0.5 x 10^9/L that is maintained for three consecutive days or a platelet count >20 x 10^9/L without a platelet transfusion in the preceding seven days. If veno-occlusive disease (VOD) occurs, the prophylaxis phase starts on the baseline date and ends on the day before the start date of rescue defibrotide. If VOD does not occur, the prophylaxis phase starts on the baseline date and ends on the date of study completion/early termination. For the subset of participants who developed VOD and received rescue defibrotide, the rescue treatment phase begins on the start date of rescue defibrotide and ends on the date of study completion/early termination.
Time Frame: Day +180 Post-HSCT
Population: Number of Participants with graft failure was assessed using the Safety Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | Defibrotide Prophylaxis | Best Supportive Care
Number analyzed (Participants) | 181 | 174
Participants
  Prophylaxis Phase | 4 | 5
  Rescue Phase | 4 | 4

36. Secondary Outcome: Number of Participants With Neutrophil Engraftment by Day +180 Post-Hematopoietic Stem Cell Transplant (HSCT)
Description: The date of neutrophil engraftment was recorded on the electronic case report form (eCRF) and is defined as the first date after HSCT of an absolute neutrophil count >0.5 x 10^9/L that is maintained for three consecutive days. The definition of "absolute neutrophil count" includes both segmented neutrophils and "bands," immature neutrophils. The number of participants with neutrophil engraftment was assessed.
Time Frame: Day +180 Post-HSCT
Population: Number of participants with neutrophil engraftment was assessed using the Safety Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | Defibrotide Prophylaxis | Best Supportive Care
Number analyzed (Participants) | 181 | 174
Participants | 156 | 162

37. Secondary Outcome: Number of Participants With Platelet Engraftment by Day +180 Post-Hematopoietic Stem Cell Transplant (HSCT)
Description: The date of platelet engraftment was recorded on the electronic case report form (eCRF) and is defined as the first date after HSCT of a platelet count >20 x 10^9/L without a platelet transfusion in the preceding seven days. The number of participants with platelet engraftment was assessed.
Time Frame: Day +180 Post-HSCT
Population: Number of Participants with platelet engraftment was assessed using the Safety Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | Defibrotide Prophylaxis | Best Supportive Care
Number analyzed (Participants) | 181 | 174
Participants | 154 | 163

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) were reported from the date of consent through Day +180 post-HSCT/Study Completion or Early Termination, or up to 4 years, 1 month.
Description: A treatment-emergent adverse event was defined as any event with onset date on or after the first dose of study treatment or any ongoing event that worsens in severity after the date of the first dose of the study treatment through the protocol-specific reporting period. Only serious adverse events considered by the investigator to be possibly related to study drug were reported more than 30 days after the last dose of the study drug. Adverse Events were assessed with the safety analysis set.
Arm/Group | Defibrotide Prophylaxis | Best Supportive Care
All-Cause Mortality (participants affected / at risk) | 35/181 | 29/174
Serious Adverse Events (participants affected / at risk) | 82/181 | 74/174
Other Adverse Events (participants affected / at risk) | 180/181 | 174/174
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Defibrotide Prophylaxis (N=181) | Best Supportive Care (N=174)
Air embolism (Vascular disorders) | 0 | 1
Capillary leak syndrome (Vascular disorders) | 1 | 0
Hypertension (Vascular disorders) | 0 | 1
Hypotension (Vascular disorders) | 3 | 2
Hypovolaemic shock (Vascular disorders) | 0 | 1
Shock (Vascular disorders) | 0 | 1
Venoocclusive disease (Vascular disorders) | 9 | 5
Acute leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Acute lymphocytic leukaemia recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Acute myeloid leukaemia recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Burkitt's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Leukaemia recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Acute graft versus host disease in intestine (Immune system disorders) | 3 | 4
Acute graft versus host disease in liver (Immune system disorders) | 0 | 1
Acute graft versus host disease in skin (Immune system disorders) | 4 | 1
Anaphylactic reaction (Immune system disorders) | 1 | 0
Cytokine release syndrome (Immune system disorders) | 1 | 0
Airway complication of anaesthesia (Injury, poisoning and procedural complications) | 0 | 1
Deep vein thrombosis postoperative (Injury, poisoning and procedural complications) | 0 | 1
Delayed engraftment (Injury, poisoning and procedural complications) | 0 | 1
Engraft failure (Injury, poisoning and procedural complications) | 1 | 0
Subarachnoid haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Subcutaneous haematoma (Injury, poisoning and procedural complications) | 0 | 1
Transplant failure (Injury, poisoning and procedural complications) | 0 | 1
Traumatic haematoma (Injury, poisoning and procedural complications) | 1 | 0
Vascular access complication (Injury, poisoning and procedural complications) | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 1
Blood bilirubin increased (Investigations) | 1 | 2
Blood creatinine increased (Investigations) | 1 | 0
Cytomegalovirus test positive (Investigations) | 1 | 1
Electrocardiogram QT prolonged (Investigations) | 1 | 0
Epstein-Barr virus test positive (Investigations) | 1 | 0
Klebsiella test positive (Investigations) | 1 | 0
Neutrophil count decreased (Investigations) | 1 | 1
Norovirus test positive (Investigations) | 0 | 1
Weight decreased (Investigations) | 1 | 0
Cardiac arrest (Cardiac disorders) | 1 | 1
Cardiac failure (Cardiac disorders) | 1 | 0
Cardio-respiratory arrest (Cardiac disorders) | 1 | 0
Pericardial effusion (Cardiac disorders) | 1 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 1
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 3 | 3
Histiocytosis haematophagic (Blood and lymphatic system disorders) | 3 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
Thrombotic microangiopathy (Blood and lymphatic system disorders) | 2 | 3
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 4 | 0
Idiopathic pneumonia syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Laryngospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pharyngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary alveolar haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 6 | 6
Respiratory tract haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Stridor (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Upper airway obstruction (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary arterial hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Cerebellar haemorrhage (Nervous system disorders) | 0 | 1
Cerebral haemorrhage (Nervous system disorders) | 1 | 1
Encephalopathy (Nervous system disorders) | 1 | 0
Haemorrhage intracranial (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 0 | 1
Leukoencephalopathy (Nervous system disorders) | 1 | 0
Nervous system disorder (Nervous system disorders) | 0 | 1
Neuralgia (Nervous system disorders) | 1 | 0
Posterior reversible encephalopathy syndrome (Nervous system disorders) | 1 | 0
Presyncope (Nervous system disorders) | 1 | 0
Seizure (Nervous system disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Anal inflammation (Gastrointestinal disorders) | 1 | 1
Colitis (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 5
Enteritis (Gastrointestinal disorders) | 1 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 3 | 0
Haematemesis (Gastrointestinal disorders) | 2 | 0
Haematochezia (Gastrointestinal disorders) | 1 | 1
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Melaena (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 1
Pneumatosis intestinalis (Gastrointestinal disorders) | 0 | 1
Stomatitis (Gastrointestinal disorders) | 1 | 3
Vomiting (Gastrointestinal disorders) | 0 | 1
Gait disturbance (Gastrointestinal disorders) | 1 | 0
General physical health deterioration (Gastrointestinal disorders) | 0 | 1
Influenza like illness (Gastrointestinal disorders) | 0 | 1
Mucosal haemorrhage (Gastrointestinal disorders) | 1 | 0
Multiple organ dysfunction syndrome (Gastrointestinal disorders) | 3 | 2
Pneumatosis (Gastrointestinal disorders) | 0 | 1
Pyrexia (Gastrointestinal disorders) | 10 | 14
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0
Hepatic failure (Hepatobiliary disorders) | 0 | 1
Venoocclusive liver disease (Hepatobiliary disorders) | 2 | 4
Acute kidney injury (Renal and urinary disorders) | 3 | 4
Anuria (Renal and urinary disorders) | 0 | 1
Cystitis haemorrhagic (Renal and urinary disorders) | 1 | 0
Nephropathy (Renal and urinary disorders) | 1 | 0
Nephropathy toxic (Renal and urinary disorders) | 0 | 1
Renal failure (Renal and urinary disorders) | 2 | 1
Renal impairment (Renal and urinary disorders) | 1 | 0
Renal injury (Renal and urinary disorders) | 0 | 1
Renal tubular dysfunction (Renal and urinary disorders) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 0
Adenovirus infection (Infections and infestations) | 1 | 2
BK virus infection (Infections and infestations) | 2 | 0
Bacterial infection (Infections and infestations) | 1 | 0
Bronchopulmonary aspergillosis (Infections and infestations) | 1 | 0
Candida sepsis (Infections and infestations) | 1 | 0
Cellulitis of male external genital organ (Infections and infestations) | 1 | 0
Clostridium difficile colitis (Infections and infestations) | 1 | 0
Croup infectious (Infections and infestations) | 1 | 0
Cystitis viral (Infections and infestations) | 1 | 1
Cytomegalovirus colitis (Infections and infestations) | 0 | 1
Cytomegalovirus infection (Infections and infestations) | 2 | 2
Cytomegalovirus viraemia (Infections and infestations) | 0 | 1
Device related infection (Infections and infestations) | 2 | 3
Device related sepsis (Infections and infestations) | 0 | 1
Epstein-Barr virus infection (Infections and infestations) | 0 | 1
Herpes zoster (Infections and infestations) | 1 | 0
Infection (Infections and infestations) | 1 | 0
Klebsiella sepsis (Infections and infestations) | 1 | 0
Meningitis (Infections and infestations) | 0 | 1
Meningoencephalitis herpetic (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 4
Pseudomonal sepsis (Infections and infestations) | 1 | 0
Respiratory tract infection (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 6 | 5
Septic shock (Infections and infestations) | 2 | 0
Skin candida (Infections and infestations) | 0 | 1
Skin infection (Infections and infestations) | 1 | 0
Staphylococcal bacteraemia (Infections and infestations) | 1 | 1
Staphylococcal sepsis (Infections and infestations) | 1 | 0
Staphylococcal skin infection (Infections and infestations) | 0 | 1
Subcutaneous abscess (Infections and infestations) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Defibrotide Prophylaxis (N=181) | Best Supportive Care (N=174)
Hypertension (Vascular disorders) | 71 (92) | 55 (80)
Hypotension (Vascular disorders) | 28 (30) | 26 (32)
Venoocclusive disease (Vascular disorders) | 8 (8) | 20 (21)
Acute graft versus host disease in intestine (Immune system disorders) | 13 (15) | 19 (19)
Acute graft versus host disease in skin (Immune system disorders) | 31 (39) | 34 (41)
Engraftment syndrome (Immune system disorders) | 14 (14) | 15 (15)
Asthenia (General disorders) | 10 (11) | 7 (7)
Chills (General disorders) | 11 (16) | 14 (16)
Face oedema (General disorders) | 10 (10) | 12 (16)
Fatigue (General disorders) | 24 (35) | 23 (28)
Malaise (General disorders) | 7 (12) | 11 (16)
Oedema peripheral (General disorders) | 27 (33) | 30 (38)
Pain (General disorders) | 22 (24) | 19 (20)
Pyrexia (General disorders) | 113 (201) | 113 (202)
Anxiety (Psychiatric disorders) | 14 (14) | 19 (20)
Depression (Psychiatric disorders) | 11 (11) | 3 (4)
Insomnia (Psychiatric disorders) | 17 (19) | 31 (35)
Infusion related reaction (Injury, poisoning and procedural complications) | 15 (20) | 12 (16)
Activated partial thromboplastin time prolonged (Investigations) | 17 (33) | 13 (33)
Alanine aminotransferase increased (Investigations) | 18 (31) | 28 (48)
Aspartate aminotransferase increased (Investigations) | 15 (31) | 28 (50)
Blood bilirubin increased (Investigations) | 26 (61) | 20 (36)
Blood creatinine increased (Investigations) | 10 (25) | 11 (16)
Cytomegalovirus test positive (Investigations) | 16 (19) | 9 (15)
International normalised ratio increased (Investigations) | 10 (22) | 12 (16)
Lymphocyte count decreased (Investigations) | 6 (13) | 10 (24)
Neutrophil count decreased (Investigations) | 19 (42) | 25 (74)
Platelet count decreased (Investigations) | 34 (168) | 43 (161)
Weight decreased (Investigations) | 22 (33) | 17 (21)
White blood cell count decreased (Investigations) | 22 (41) | 17 (68)
Sinus tachycardia (Cardiac disorders) | 37 (47) | 24 (30)
Cough (Respiratory, thoracic and mediastinal disorders) | 24 (29) | 23 (26)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 12 (15) | 11 (11)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 41 (52) | 46 (68)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 13 (15) | 10 (10)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 10 (13) | 4 (4)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 20 (21) | 20 (26)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 15 (16) | 7 (9)
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 10 (10) | 8 (8)
Anaemia (Blood and lymphatic system disorders) | 50 (163) | 52 (158)
Febrile neutropenia (Blood and lymphatic system disorders) | 52 (57) | 59 (70)
Leukopenia (Blood and lymphatic system disorders) | 5 (9) | 10 (22)
Neutropenia (Blood and lymphatic system disorders) | 31 (52) | 27 (44)
Thrombocytopenia (Blood and lymphatic system disorders) | 31 (56) | 27 (77)
Headache (Nervous system disorders) | 50 (77) | 36 (60)
Abdominal distension (Gastrointestinal disorders) | 17 (21) | 4 (4)
Abdominal pain (Gastrointestinal disorders) | 57 (87) | 48 (70)
Abdominal pain upper (Gastrointestinal disorders) | 12 (16) | 11 (11)
Constipation (Gastrointestinal disorders) | 40 (44) | 39 (40)
Diarrhoea (Gastrointestinal disorders) | 110 (176) | 108 (178)
Haemorrhoids (Gastrointestinal disorders) | 12 (14) | 13 (15)
Nausea (Gastrointestinal disorders) | 109 (166) | 101 (149)
Oral pain (Gastrointestinal disorders) | 13 (14) | 8 (10)
Proctalgia (Gastrointestinal disorders) | 7 (8) | 9 (11)
Stomatitis (Gastrointestinal disorders) | 105 (167) | 114 (188)
Vomiting (Gastrointestinal disorders) | 106 (208) | 91 (179)
Acute kidney injury (Renal and urinary disorders) | 8 (11) | 14 (18)
Haematuria (Renal and urinary disorders) | 21 (23) | 13 (17)
Dry skin (Skin and subcutaneous tissue disorders) | 21 (26) | 11 (13)
Erythema (Skin and subcutaneous tissue disorders) | 13 (15) | 14 (16)
Pruritus (Skin and subcutaneous tissue disorders) | 13 (14) | 24 (26)
Pruritus generalised (Skin and subcutaneous tissue disorders) | 13 (17) | 11 (13)
Rash (Skin and subcutaneous tissue disorders) | 32 (43) | 20 (26)
Rash generalised (Skin and subcutaneous tissue disorders) | 12 (13) | 6 (8)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 13 (15) | 12 (16)
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 (9) | 10 (11)
Back pain (Musculoskeletal and connective tissue disorders) | 18 (20) | 8 (8)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 19 (25) | 15 (18)
Decreased appetite (Metabolism and nutrition disorders) | 51 (75) | 51 (72)
Fluid overload (Metabolism and nutrition disorders) | 13 (16) | 8 (12)
Fluid retention (Metabolism and nutrition disorders) | 14 (15) | 16 (18)
Hyperglycaemia (Metabolism and nutrition disorders) | 22 (31) | 17 (35)
Hyperkalaemia (Metabolism and nutrition disorders) | 12 (16) | 12 (18)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 29 (60) | 23 (55)
Hypocalcaemia (Metabolism and nutrition disorders) | 19 (28) | 24 (48)
Hypokalaemia (Metabolism and nutrition disorders) | 75 (114) | 63 (111)
Hypomagnesaemia (Metabolism and nutrition disorders) | 71 (123) | 59 (123)
Hyponatraemia (Metabolism and nutrition disorders) | 17 (24) | 13 (19)
Hypophosphataemia (Metabolism and nutrition disorders) | 20 (34) | 23 (40)
Cytomegalovirus infection (Infections and infestations) | 26 (29) | 23 (24)
Cytomegalovirus viraemia (Infections and infestations) | 6 (7) | 9 (9)
Device related infection (Infections and infestations) | 15 (17) | 9 (9)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-08-20): https://cdn.clinicaltrials.gov/large-docs/07/NCT02851407/Prot_000.pdf
  • Statistical Analysis Plan (2020-11-24): https://cdn.clinicaltrials.gov/large-docs/07/NCT02851407/SAP_001.pdf